CLINICAL TRIAL: NCT01420419
Title: A Randomized Controlled Trial Evaluating Lanolin for the Treatment of Nipple Pain Among Breastfeeding Women
Brief Title: Evaluating Lanolin for the Treatment of Nipple Pain Among Breastfeeding Women
Acronym: LanP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Cindy-Lee Dennis, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26044
Record Dates: First submitted 2011-03-29; First posted 2011-08-19 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Pain
Keywords: nipple pain; breastfeeding; nipple damage; lanolin; clinical trial
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Lanolin; Hospitals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lanolin (Experimental): Pea sized amount of lanolin to be applied to nipple and areola after every breast feed (approximately every 2-3 hours), until pain is completely resolved for a maximum of 7 days
  Interventions: Other: Lanolin
- Standard postpartum nursing care (Other): Women in standard care control group may receive any other nursing intervention to manage their nipple pain, including (but not limited to): recommending application of expressed breast milk, analgesics (such as acetaminophen or ibuprofen), breast shells, air drying, changing position / latch, cold or warm compresses
  Interventions: Other: Standard (usual) in-hospital and community postpartum care

INTERVENTIONS:
Other: Lanolin — Pea-sized amount of lanolin applied to each nipple after every breastfeeding session (approximately 8-12 times daily) until complete resolution of nipple pain and damage for a maximum of 7 days.
  Arms: Lanolin
Other: Standard (usual) in-hospital and community postpartum care — Women randomized to standard care will not receive lanolin or information regarding how to use lanolin. In-hospital standard care may include any of the following pain management measures at the recommendation / discretion of the participant's health care provider, or based on the patient's personal preference: analgesics (such as ibuprofen or acetaminophen); application of cold or warm compresses; application of ice packs; use of breast shields; air drying the nipples; or applying expressed breast milk.
  Arms: Standard postpartum nursing care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of lanolin for the treatment of painful/damaged nipples among breastfeeding women, and to evaluate if the use of lanolin has an effect on breastfeeding outcomes such as duration and exclusivity.

ELIGIBILITY:
Inclusion Criteria:

* Maternal complaint of nipple pain with any sign of nipple trauma to one or both nipples, such as blistering, crusting, redness, bleeding, swelling, cracking, discoloration or peeling.
* Infant delivered at, or greater than 37 weeks gestation.
* Singleton birth.
* Speaks and understands English.
* Access to telephone.

Exclusion Criteria:

* Infant not expected to be discharged home with mother.
* Infant with congenital abnormalities that would impair breastfeeding.
* Maternal allergy to lanolin.
* Maternal health conditions that may interfere with breastfeeding (physical or mental illness) as determined by hospital staff.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Nipple pain severity | 4 days post randomization
  Measured with a 10-point numeric rating scale (NRS)

SECONDARY OUTCOMES:
Breastfeeding duration | 4 and 12 weeks postpartum
  Measured by asking women the last time their infant was breastfed. Breastfeeding duration will be calculated as the difference between the infant's date of birth, and the last day (date) the infant was breastfed.
Breastfeeding exclusivity | 4 and 12 weeks postpartum
  Measured with Labbok & Krasovek's framework for breastfeeding definition (Studies in Family Planning, 1990;21(4),226-230)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy-Lee Dennis, PhD, Principal Investigator — University of Toronto
Locations (1):
- Postpartum Unit St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada